CLINICAL TRIAL: NCT00622063
Title: An Extension Study for Patients Previously Treated With ARQ 501
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 501-115
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Cancer
Keywords: cancer, solid tumor
MeSH Terms: conditions — Neoplasms | interventions — beta-lapachone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ARQ 501 — Treatment with ARQ 501 or ARQ 501 as combination therapy at the dose and regimen previously received

SUMMARY:
To provide ongoing treatment with ARQ 501 for patients who have benefited from prior treatment with ARQ 501

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Has previous participated in a clinical trial with ARQ 501 and is eligible for continued treatment

Exclusion Criteria:

* Have not received previous treatment with ARQ 501 under a treatment protocol
* Uncontrolled intercurrent illness, uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To provide ongoing treatment with ARQ 501 for patients who have benefited from prior treatment with ARQ 501 | No time frame

SECONDARY OUTCOMES:
To collect additional safety and tolerability information for ARQ 501 treatment | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Neil Nathan Senzer, MD, Principal Investigator — Mary Crowley Medical Research Center
Locations (1):
- Mary Crowley Medical Research Center, Dallas, Texas, United States